CLINICAL TRIAL: NCT04023292
Title: Comparative Study for the Degree of Biological Changes After Short-term 2 Weeks and 4 Weeks Preoperative Endocrine Therapy in Luminal Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Shicheng Su, Director of Shuhua Breast Cancer Research Center of Sun Yat-sen Memorial Hospital, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-KY-051; ChiCTR1900024427 (Registry Identifier: Chinese Clinical Trial Registry)
Record Dates: First submitted 2019-07-15; First posted 2019-07-17 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Breast Neoplasms
Keywords: Hormone receptors-positive breast neoplasms; preoperative endocrine therapy; Ki-67
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen; Letrozole; Anastrozole; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (2 weeks preoperative endocrine therapy)) (Experimental): Patients receive endocrine therapy before surgery for 2 weeks. Choice of endocrine therapy is according to guidelines and centre policy.
  Interventions: Drug: Endocrine therapy
- Arm II (4 weeks preoperative endocrine therapy) (Active Comparator): Patients receive endocrine therapy before surgery for 4 weeks. Choice of endocrine therapy is according to guidelines and centre policy.
  Interventions: Drug: Endocrine therapy

INTERVENTIONS:
Drug: Endocrine therapy — Use before surgery for 2 weeks. Choice of endocrine therapy is according to guidelines and centre policy.
  Other Names: tamoxifen, Letrozole, Anastrazole, Exemestane, etc.
  Arms: Arm I (2 weeks preoperative endocrine therapy))
Drug: Endocrine therapy — Use before surgery for 4 weeks. Choice of endocrine therapy is according to guidelines and centre policy.
  Other Names: tamoxifen, Letrozole, Anastrazole, Exemestane, etc.
  Arms: Arm II (4 weeks preoperative endocrine therapy)

SUMMARY:
RATIONALE: Estrogen can promote proliferation of tumor cells in hormone receptors (HR)-positive breast cancer. The standard therapy of Luminal subtypes is endocrine therapy, which can influence proliferation of tumor cells by blocking the use of estrogen by cancer cells or lowering the amount of estrogen the body makes. Thus, markers of proliferation are candidate markers of efficacy after short-term (e.g., 2 weeks or 4 weeks) preoperative hormone therapy. Ki-67 is most commonly used among these markers. In contrast to the absolute value, the degree of Ki-67 changes which consider the baseline values would be better to reflect the sensitivity of therapy. It is not yet known whether the degree of Ki-67 changes after 2 weeks or 4 weeks presurgery endocrine therapy is different and which interval is more suitable to assess therapy sensitivity.

PURPOSE: This randomized phase II trial is studying to compare the degree of Ki-67 changes after 2 weeks or 4 weeks preoperative endocrine therapy and to determine a more appropriate interval to assess hormone therapy sensitivity in women who are undergoing surgery for HR-positive, Human epidermal growth factor receptor 2 (HER2)-negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Signed the informed consent.
2. Female aged between 18 and 70 years.
3. Pathologically diagnosed operable invasive breast cancer meeting the following criterias:

   * Hormone receptor (HR)-positive: pathologically diagnosed estrogen receptor (ER)-positive and/or progesterone receptor (PR)-positive;
   * Human epidermal growth factor receptor 2 (HER2)-negative: FISH or immunohistochemistry (IHC).
4. WHO Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
5. Newly diagnosed breast cancer.
6. The important organ functions meet the following criterias:

   * WBC >=3.0 x 10^9/L; Neutrophilic granulocytes >=1.5×10^9/L; Platelet >=100 x 10^9/L; Hb >=9 g/dL;
   * Total bilirubin no more than 1.5 times the normal upper limit (ULN); AST and ALT no more than 1.5 times ULN; AKP no more than 2.5 times ULN;
   * Serum creatinine no more than 1.5 times ULN or Clearance rate of creatinine >= 60ml/min;
   * Thyroid stimulating hormone (TSH) <= ULN (T3, T4 levels need to be detected simultaneously if abnormalities, the patient can be included if T3, T4 levels is normal);
   * LVEF basement >= 50%.
7. Able to swallow tablets.
8. Pregnancy test (serum or urine HCG test within 72h before enrollment) must be negative in non-surgical sterilization or women of childbearing age, must be not for the nursing and be willing to take non-pharmacological contraception during treatment (such as intrauterine device, condom, etc).

Exclusion Criteria:

1. Evidence of distant metastasis.
2. Bilateral or multiple unilateral breast tumors with different histological characteristics (such as ER/PR/HER2 status, tumor grade or type, etc).
3. Any invasive malignancy diagnosed within previous 5 years (other than successfully treated cervical carcinoma in situ, skin basal cell carcinoma or cutaneous squamous cell carcinoma).
4. Prior radiotherapy, chemotherapy, endocrine therapy, targeted therapy etc.
5. Concurrent use of HRT or any other estrogen-containing medication (including vaginal estrogens) within 4 weeks.
6. Prior use of estrogen implants.
7. Prior use of high-dose systemic corticosteroids (except as antiemetic treatment), immunotherapy, or biological response modifiers (e.g., interferon, etc).
8. Use of an unlicensed or other investigational drug within 4 weeks.
9. Any severe comorbidities, inability to give informed consent or unavailability for follow-up, including but not limited to any of the following:

   * Heart failure above NYHA class 2 level; high-risk uncontrollable arrhythmia; unstable angina pectoris; myocardial infarction within 1 year; valvular heart disease with clinically significance or requiring intervention.
   * Chronic obstructive pulmonary disease requires treatment.
   * Chronic liver disease (cirrhosis, chronic active hepatitis, etc).
   * Cerebrovascular accident occurred within 6 months.
   * Severe epilepsy or central nervous system diseases.
   * Hypertension which cannot be well controlled by antihypertensive drugs.
   * Abnormal coagulation, bleeding tendency, or receiving thrombolysis or anticoagulant therapy.
   * Chronic renal insufficiency.
   * Active infection.
   * Psychiatric disability, etc.
10. Pregnant or nursing females.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Percentage Change From Pre-treatment to Post-treatment in Ki-67 Labelling Index | 2 weeks or 4 weeks endocrine treatment before surgery
  Ki-67 labelling index is calculated as the percentage of cells with Ki-67-positive nuclear immunostaining as measured by immunohistochemistry (IHC). Range 0-100. Percentage change from pre-treatment to post-treatment=[(Ki-67post - Ki-67pre)/Ki-67pre]x100%

SECONDARY OUTCOMES:
Disease Free Survival (DFS) | 5 years post-randomisation
Overall Survival (OS) | 5 years post-randomisation

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong, China